## Statistical Analysis Plan

Ronald Seidel, MD

Eduard Barbakov, MD

HELIOS Medical Center Schwerin

Department for Anesthesiology

Wismarsche Strasse 393-7, DE-19049 Schwerin, Germany

## Title

Surgical treatment of proximal femoral fractures under peripheral regional anesthesia. A prospective pilot study.

ID: A 2018-0237 NCT: 04005404

**Final Version** 

Date 29.06.2019

## **Statistical Analysis Plan**

The metric parameters are described by mean value (Mw) and standard deviation (Sd). The Mann-Whitney U test tests whether the two groups differ in the distribution of the parameter. If the p-value of the test is less than the selected significance level (0.05), then the groups differ significantly in terms of distribution.

Categorical parameters (0/1) are described by the exact Fisher test. The exact Fisher test examines whether each parameter is independent of its membership in a group. If the p-value of the test is less than the selected significance level (0.05), then there is a significant dependence. The two groups then differ significantly with respect to the selected parameter.

The incidence of adverse events in the two groups is described with odds ratios (95% confidence interval).

Statistical analyses were performed bilaterally, using GraphPad PRISM 8.0 (GraphPad Software Inc., San Diego, CA, USA).